CLINICAL TRIAL: NCT00799929
Title: Efficiency and Patient Satisfaction of Two Different IVF Protocols.
Brief Title: IVF Clinical Trial of Two Different Treatment Protocols.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New Hope Fertility Center (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JZ-09-08; NHFC
Record Dates: First submitted 2008-11-26; First posted 2008-12-01 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Infertility
Keywords: IVF Research Study; Infertility Sudy; in vitro fertilization; Mini IVF; Conventional IVF
MeSH Terms: conditions — Infertility | interventions — Fertilization in Vitro

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARM A - Mini IVF (Active Comparator): The Mini IVF method entails pre-treatment with oral contraceptive pills. Ovarian stimulation is achieved using an oral anti-estrogen in conjunction with injections of gonadotropin (225IU-600IU per cycle), with initial dose of 75IU-150IU per injection. Ovulation is induced by a GnRH (gonadotropin-releasing hormone) agonist nasal spray/hCG (human chorionic gonadotropin) injection. Retrieved oocytes following in vitro fertilization (IVF/ICSI) are cultured to the blastocyst stage. Blastocyst stage embryos are vitrified using the CryoTop method. No fresh embryo transfer is conducted. Subsequently, SET of a thawed blastocyst is performed in a natural cycle/HRT that does not involve ovarian stimulation. SETs are conducted until pregnancy is achieved or all vitrified blastocysts have been used.
  Interventions: Other: in vitro fertilization (IVF/ICSI)
- Arm B - Conventional IVF (Active Comparator): The standard IVF method entails pre-treatment with a GnRH analog injections in the midluteal phase. Controlled ovarian hyperstimulation is achieved with injections of gonadotropin (150IU-300IU/day). Ovulation is induced by hCG injection and retrieved oocytes following in vitro fertilization (IVF/ICSI) are cultured to the blastocyst stage. If this occurs on day 5, then fresh SET/DET (single embryo transfer/double embryo transfer) is performed. Remaining blastocysts are cryopreserved and transferred in subsequent natural cycles/HRT (hormone replacement therapy) that does not involve ovarian stimulation.
  Interventions: Other: in vitro fertilization (IVF/ICSI)

INTERVENTIONS:
Other: in vitro fertilization (IVF/ICSI)

SUMMARY:
The purpose of this study is to compare two different in vitro fertilization (IVF) treatments: conventional IVF protocol and minimal stimulation IVF protocol, in terms of success rates, stress of treatment, drug-related side effects, multiple pregnancies and cost of treatment.

DETAILED DESCRIPTION:
A random population of 564 sub-fertile women or couples with a female between ages of 18 and 38 years and a desire to undergo their first IVF cycle will be included in this outpatient clinical trial. The participation in this study will be approximately six months with a total of 20 to 25 visits. After successful completion of the pre-screening tests participants are randomized into one of the two arms of the study: Arm A - mini IVF protocol, and Arm B - conventional IVF protocol.

ELIGIBILITY:
Inclusion criteria:

* Valid indication for IVF treatment
* First IVF attempt
* Female age between 18 and 38 years
* Male partner 18 years of age or older
* Both partners STD free
* Must be able to understand that they may NOT become pregnant

Exclusion criteria:

* Not willing or able to sign the consent form
* Pre-existing medical condition preventing/interfering with IVF treatment
* Abnormal IVF screening tests, which includes Complete Blood Count, Varicella titer, Rubella titer, PAP smear, Syphilis, HIV 1&2, Hepatitis B, Hepatitis C, Chlamydia, and Gonorrhea
* Abnormal pap smear
* Body Mass Index (BMI) falls below 18.5 or above 32.0
* Female participant with irregular menstrual cycles

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 564 (Actual)
Dates: Start 2008-12; Primary Completion 2014-05 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Primary outcome parameter: Live birth | 4 Years

SECONDARY OUTCOMES:
Secondary outcome parameters: Biochemical pregnancy, Clinical pregnancy, Ongoing pregnancy, Multiple pregnancy rate, Miscarriage rate, Fertilization rate, Number of oocytes, Number of embryos | 4 Years

CONTACTS AND LOCATIONS:
Overall Officials: John J Zhang, MD, MSc, PhD, Principal Investigator — New Hope Fertility Center
Locations (1):
- New Hope Fertility Center, New York, New York, United States

REFERENCES:
- [Derived] Zhang JJ, Yang M, Merhi Z. Efficiency of metaphase II oocytes following minimal/mild ovarian stimulation in vitro fertilization. Fertil Res Pract. 2016 Sep 1;2:2. doi: 10.1186/s40738-016-0025-6. eCollection 2016. PMID 28620528